CLINICAL TRIAL: NCT07402993
Title: DASH Diet and Cardiometabolic Risk in Parkinson's Disease: Lower Triglycerides and AIP With Higher Adherence
Brief Title: DASH Diet, Triglycerides and AIP in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Nurefşan KONYALIGİL ÖZTÜRK, Assist. Prof. Dr, Abant Izzet Baysal University
Other Study IDs: AIBU-BD-NKÖ-04
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease
Keywords: Cardiovascular risk; DASH diet; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Parkinson's disease: This cohort includes adult participants diagnosed with Parkinson's disease. No control group is included.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
Participants who agreed to participate in the study were informed about the purpose of the research and obtained their consent to participate in the study using an informed consent form. The study was conducted on 70 patients with Parkinson's disease. Participants who volunteered to participate in the study were given a questionnaire form containing sociodemographic characteristics. In addition, participants' anthropometric measurements (body weight, height, waist and hip circumference, Body Mass Index (BMI)), biochemical parameters (fasting blood glucose, HbA1c, triglycerides, LDL cholesterol, triglycerides, total cholesterol, C-reactive protein (CRP), albumin, and hematology markers (hemoglobin (Hb), hematocrit (Htc), leukocytes and platelets, lymphocytes) and serum vitamin D, folic acid, vitamin B12) and nutritional status (food consumption frequency, DASH diet compliance) were obtained. New cardiovascular risk markers such as neutrophil/lymphocyte ratio (NLR), monocyte HDL ratio (MHR), and plasma atherogenic index (PAI) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 19 years of age
* Individuals who are literate
* Individuals diagnosed with Parkinson's Disease

Exclusion Criteria:

* Individuals who have had an acute infection or inflammatory disease within the past month
* Individuals with chronic infectious or inflammatory diseases
* Individuals with cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was designed as a cross-sectional descriptive study. The study included patients who presented to the Neurology Outpatient Clinic at BAİBÜ İzzet Baysal Education and Research Hospital and diagnosed with Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire Form | 6 months
  Sociodemographic characteristics of the individuals (age, constipation status, presence of comorbidities, gender, smoking and alcohol use) were questioned.
Body weight (BW) | 6 months
  BW was measured using a calibrated digital scale placed on a flat, tiled surface. The scale was sensitive to 100 grams.
Height | 6 months
  Height was measured using a stadiometer with the participant's head positioned in the Frankfort plane and feet placed together.
Waist Circumference (WC) | 6 months
  WC was measured at the midpoint between the lowest rib and the iliac crest (cristal point) using a flexible measuring tape.
Hip Circumference (HC) | 6 months
  HC was measured at the widest point of the hips using a flexible measuring tape.
Body Mass Index (BMI) | 6 months
  BMI was calculated by dividing body weight (in kilograms) by the square of height (in meters): BMI = weight (kg) / height² (m²).
Fasting Blood Glucose | 6 months
  Fasting blood glucose was measured using standard laboratory techniques during routine outpatient visits.
Triglycerides | 6 months
  Triglyceride levels were measured via fasting blood samples analyzed in the outpatient clinic laboratory.
LDL-Cholesterol | 6 months
  LDL-cholesterol was measured from fasting serum samples using standard enzymatic colorimetric methods.
HDL-Cholesterol | 6 months
  HDL-cholesterol was measured from fasting serum samples using standard enzymatic colorimetric methods.
C-Reactive Protein (CRP) | 6 months
  CRP levels were measured using routine laboratory procedures in outpatient visits.
Vitamin D | 6 months
  Serum vitamin D (25(OH)D) levels were assessed using chemiluminescence immunoassay methods in the outpatient clinic laboratory.
Folic Acid | 6 months
  Serum folic acid levels were measured using standard automated immunoassay techniques.immunoassay methods in the outpatient clinic laboratory.
Vitamin B12 | 6 months
  Serum vitamin B12 concentrations were measured using automated chemiluminescent immunoassay.immunoassay methods in the outpatient clinic laboratory.
Atherogenic Index of Plasma (AIP) | 6 months
  AIP is a logarithmically transformed ratio of plasma triglycerides to high-density lipoprotein cholesterol [log₁₀(TG/HDL-C)], and it is used as a surrogate marker of atherogenicity and cardiovascular risk.
Monocyte-to-High-Density Lipoprotein Cholesterol Ratio | 6 months
  A biomarker reflecting the balance between inflammatory status (monocytes) and anti-atherogenic lipid components (HDL-C); it has been proposed as an indicator of systemic inflammation and cardiovascular risk.
Total Cholesterol-to-High-Density Lipoprotein Cholesterol Ratio | 6 months
  A widely used index of atherogenic risk, representing the balance between total cholesterol and protective HDL-C, with higher values indicating increased cardiovascular risk.
Neutrophil-to-Lymphocyte Ratio (NLR) | 6 months
  A systemic inflammatory marker calculated as the ratio of neutrophils to lymphocytes, commonly used to assess inflammatory status and immune response.
Food consumption frequency | 6 months
  Participants were asked about the foods they consumed in the past month from seven groups, including five basic food groups (meat and meat products, milk and dairy products, bread and grains, vegetables and fruits, sugars and fats), beverages, and fast food. Participants were asked how often and in what quantities they consumed these foods using eight options: "every meal," "every day," "5-6 days a week," "3-4 days a week," "1-2 days a week," "once every 15 days," "once a month," and "never." In evaluating food consumption records, responses regarding food consumption frequency were calculated using food consumption frequency. The amounts of food and beverages consumed were multiplied by "3" for "every meal," '1' for "every day," "0.7855" for "5-6 times a week," "0.498" for "3-4 times a week," "0.2145" for "1-2 times a week," "0.067" for "once every 15 days," and "0.033" for "once a month" to obtain the daily average amounts.
Food consumption record | 6 months
  A single-day food consumption record was obtained using the 24-hour recall method to determine participants' food consumption patterns. The Food and Nutrition Photo Catalog was used to estimate portions to ensure that the amounts of food consumed were assessed accurately and reliably. Based on these records, daily energy and nutrient intakes were calculated using the Nutrition Information System (BEBİS) software, based on the type and amount of food consumed by individuals in the last 24 hours.
DASH diet compliance | 6 months
  Individuals' DASH diet compliance scores were calculated based on their food consumption frequency after their energy requirements were calculated. The highest possible score on the DASH diet compliance scale is 8.0. A score of 4.5 or above is considered 'high compliance', while a score below 4.5 is considered 'low compliance'.

CONTACTS AND LOCATIONS:
Overall Officials: Nurefşan Konyalıgil Öztürk, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Bolu, Turkey (Türkiye)